CLINICAL TRIAL: NCT01852084
Title: To Evaluate the Safety and Effectiveness of the EnVista® One-Piece Hydrophobic Acrylic Toric IOL Designed to Reduce the Effects of Preoperative Corneal Astigmatism on Postoperative Refraction Following Cataract Surgery
Brief Title: Hydrophobic Acrylic Toric IOL Designed to Reduce the Effects of Preoperative Corneal Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 761
Record Dates: First submitted 2013-05-09; First posted 2013-05-13 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Intervention Model Description: A Prospective, Multicenter Clinical Trial to Evaluate the Safety and Effectiveness
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- enVista® One-Piece Hydrophobic Acrylic Toric IOL (Experimental): Toric cylinder power of either 1.25 diopters (D), 2.00 D, or 2.75 D
  Interventions: Device: enVista® One-Piece Hydrophobic Acrylic Toric IOL
- enVista control lens (Experimental): Spherical control lens
  Interventions: Device: enVista control lens

INTERVENTIONS:
Device: enVista® One-Piece Hydrophobic Acrylic Toric IOL — Test lens having a toric cylinder power of either 1.25 diopters (D), 2.00 D, or 2.75 D
  Arms: enVista® One-Piece Hydrophobic Acrylic Toric IOL
Device: enVista control lens — Spherical Control lens
  Arms: enVista control lens

SUMMARY:
The investigational enVista IOL, Model MX60Tis equipped with toric optics and axis marks on the posterior surface to minimize the possibility of surgically induced astigmatism.

DETAILED DESCRIPTION:
The investigational enVista Toric IOL, Model MX60T, and the currently approved Model MX60, are identical with the exception of the addition of toric optics and axis marks on the posterior optic surface for the correction of astigmatism on the Model MX60T. Both lenses have an aspheric biconvex optic with a modified C haptic monoblock, single-piece design. The design and material of both the MX60 and MX60T allow them to be folded and inserted through small incisions to minimize the possibility of surgically induced astigmatism (SIA).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinically significant cataract in the study eye that is considered amenable to treatment with standard phacoemulsification cataract extraction.
* Subjects must require a lens power from 16.0 D to 27.0 D in the study eye.
* Subjects must be willing to discontinue contact lens wear for the duration of the study and, demonstrate stability prior to biometry and surgery in the study eye.
* Subjects must have a best corrected distance visual acuity (BCDVA) projected to be better than 20/30 after toric IOL implantation in the study eye.
* Subjects must have predicted postoperative corneal astigmatism between 0.90D and 2.40D in the study eye, as determined by the Toric Calculator.
* Subjects must have a minimum preoperative corneal astigmatism of 0.90 D in the study eye.
* Subjects must have a dilated preoperative pupil size greater than or equal to 5.0 mm in the study eye.

Exclusion Criteria:

* Subjects who have had previous intraocular or corneal surgery in the study eye.
* Subjects with any clinically significant ocular pathology which would be expected to reduce potential BCDVA to 20/30 or worse in the study eye during the course of the study.
* Subjects with any anterior segment pathology in the study eye likely to increase the risk of complications from phacoemulsification cataract surgery.
* Subjects with associated ocular conditions which could affect the stability of the IOL in the study eye.
* Subjects with a traumatic cataract in the study eye.
* Subjects with uncontrolled glaucoma in the study eye.
* Subjects with clinically significant irregular corneal astigmatism in the study eye, as determined by the medical judgment of the Investigator.
* Subjects with clinically significant corneal pathology potentially affecting topography of either eye.
* Subjects with any ocular condition that could prevent the possibility of a visual outcome better than 20/30 in the study eye.
* Subjects with a difference of greater than 0.50D of corneal astigmatism as measured with the IOL Master and the topographer in the study eye using vector analysis.
* Subjects with an anterior chamber depth <2mm in the study eye.
* Subjects with potential BCDVA of 20/200 or worse in the fellow eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2013-03-06 (Actual); Primary Completion 2016-07-18 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Packer, MD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Control IOL: Control IOL - Spherical control lens
- Toric IOL1.25 D: Toric IOL1.25 D - Toric cylinder power of 1.25 diopters (D)
- Toric IOL 2.00 D: Toric IOL 2.00 D - - Toric cylinder power of 2.00 diopters (D)
- Toric IOL 2.75 D: Toric IOL 2.75 D - Toric cylinder power of 2.75 diopters (D)
Period: Overall Study
Arm/Group | Control IOL | Toric IOL1.25 D | Toric IOL 2.00 D | Toric IOL 2.75 D
Started | 79 | 80 | 20 | 12
Completed | 79 | 80 | 18 | 12
Not Completed | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control IOL | Toric IOL1.25 D | Toric IOL 2.00 D | Toric IOL 2.75 D | Total
Number analyzed (Participants) | 79 | 80 | 20 | 12 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (8.6) | 71.1 (8.8) | 68.7 (9.1) | 69.6 (8.8) | 70.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 49 | 8 | 9 | 102
  Male | 43 | 31 | 12 | 3 | 89

OUTCOME MEASURES:

1. Primary Outcome: Mean Dioptric Change in Cylinder
Description: Dioptric change in cylinder from the preoperative keratometric cylinder magnitude to postoperative manifest refraction cylinder magnitude (referenced to the corneal plane).
Time Frame: Baseline, Final Visit (scheduled within window: days 120-180)
Population: Evaluable participants at the specified timepoint are included in the analysis.
Measure: Mean (Standard Deviation); unit: diopter
Arm/Group | Control IOL | Toric IOL1.25 D | Toric IOL 2.00 D | Toric IOL 2.75 D
Number analyzed (Participants) | 78 | 80 | 18 | 12
diopter | -0.479 (0.665) | -0.865 (0.487) | -1.413 (0.532) | -1.944 (0.327)

2. Primary Outcome: Percentage of Participants With Intraocular Lens (IOL) Rotation of Less Than or Equal to Five Degrees
Description: Intraocular Lens (IOL) rotation of less than or equal to five degrees between Forms 3 (scheduled within window: days 30-60) and final visit (scheduled within window: days 120-180).
Time Frame: Form 3 Visit (window: days 30-60), Final Visit (window: days 120-180)
Population: The measure was not assessed for the control IOL. Evaluable participants at the specified timepoint are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Control IOL | Toric IOL1.25 D | Toric IOL 2.00 D | Toric IOL 2.75 D
Number analyzed (Participants) | 0 | 74 | 15 | 12
Participants |  | 74 | 15 | 12

3. Primary Outcome: Mean Best-corrected Distance Visual Acuity (BCDVA) at Final Visit
Description: Best-corrected distance visual acuity (BCDVA) at Final Visit, expressed as logarithm of the minimum angle of resolution (logMAR). Corrected means spectacle corrected. Visual acuity (VA) was reported as letters read correctly, and the letters read were converted to logarithm of the minimum angle of resolution (logMAR) acuity. The participant read rows of letters on a standard LogMAR chart until the participant misses 3 letters on a row with 5 letters. The total number of correct letters were recorded. A decrease in the number of correct letters indicates a decrease in visual acuity.
Time Frame: Final Visit (scheduled within window: days 120-180)
Population: Evaluable participants at the specified timepoint are included in the analysis.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control IOL | Toric IOL1.25 D | Toric IOL 2.00 D | Toric IOL 2.75 D
Number analyzed (Participants) | 78 | 80 | 18 | 12
logMAR | 0.01 (0.09) | 0.00 (0.09) | 0.05 (0.10) | -0.01 (0.09)

4. Primary Outcome: Percentage of Participants With Reduction in Cylinder Within 0.50 Diopter (D) and Within 1.00 D of Intended.
Time Frame: Final Visit (scheduled within window: days 120-180)
Population: Evaluable participants at the specified timepoint are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Control IOL | Toric IOL1.25 D | Toric IOL 2.00 D | Toric IOL 2.75 D
Number analyzed (Participants) | 78 | 80 | 18 | 12
Participants
  Within 0.50 D of intended | 27 | 43 | 12 | 8
  Within 1.00 D of intended | 45 | 71 | 17 | 12

5. Secondary Outcome: Mean Uncorrected Distance Visual Acuity (UCDVA) at Final Visit
Description: Uncorrected distance visual acuity (UCDVA), expressed as logarithm of the minimum angle of resolution (logMAR). Uncorrected means not spectacle-corrected. Visual acuity (VA) was reported as letters read correctly, and the letters read were converted to logarithm of the minimum angle of resolution (logMAR) acuity. The participant read rows of letters on a standard LogMAR chart until the participant misses 3 letters on a row with 5 letters. The total number of correct letters were recorded. A decrease in the number of correct letters indicates a decrease in visual acuity.
Time Frame: Final Visit (scheduled within window: days 120-180)
Population: Evaluable participants at the specified timepoint are included in the analysis.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control IOL | Toric IOL1.25 D | Toric IOL 2.00 D | Toric IOL 2.75 D
Number analyzed (Participants) | 78 | 80 | 18 | 12
logMAR | 0.19 (0.16) | 0.11 (0.14) | 0.12 (0.11) | 0.13 (0.18)

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | Control IOL | Toric IOL1.25 D | Toric IOL 2.00 D | Toric IOL 2.75 D
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/80 | 0/20 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/79 | 2/80 | 1/20 | 0/12
Other Adverse Events (participants affected / at risk) | 38/79 | 39/80 | 7/20 | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control IOL (N=79) | Toric IOL1.25 D (N=80) | Toric IOL 2.00 D (N=20) | Toric IOL 2.75 D (N=12)
Epiretinal membrane (Eye disorders) | 0 | 0 | 1 | 0
IOL tilt (Eye disorders) | 0 | 1 | 0 | 0
Anterior lens vault (Eye disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control IOL (N=79) | Toric IOL1.25 D (N=80) | Toric IOL 2.00 D (N=20) | Toric IOL 2.75 D (N=12)
Corneal edema (Eye disorders) | 15 | 18 | 3 | 0
Anterior chamber cell (Eye disorders) | 17 | 15 | 1 | 1
Anterior chamber flare (Eye disorders) | 4 | 3 | 1 | 1
Punctate keratosis (Eye disorders) | 6 | 5 | 0 | 0
Visual acuity reduced (Eye disorders) | 7 | 2 | 1 | 1
Dry eye (Eye disorders) | 1 | 1 | 2 | 0
Diplopia (Eye disorders) | 0 | 1 | 1 | 0
Trichiasis (Eye disorders) | 0 | 1 | 1 | 0
Maculopathy (Eye disorders) | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 3 | 5 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.